CLINICAL TRIAL: NCT01138228
Title: Validation of Vue Tek Digital Vein Viewing Device
Brief Title: Does the VTS1000 Infra Red Vein Imager Allow Better Identification of Veins Than Normal Eyesight?
Acronym: VFvalidation
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Vue Tek Scientific (Unknown)
Responsible Party: Franco Resta-Flarer, M.D., St. Luke's Roosevelt Hospitals
Other Study IDs: VF Validation
Record Dates: First submitted 2010-03-03; First posted 2010-06-07 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-02

CONDITIONS: Vision
Keywords: intravenous cannulation; vein identification; vascular identification; vein cannulation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal vision: This within-subjects design is counter balanced for order. Each operator sees the subject's arm either initially with the normal eye or with the device, then repeats with the second condition (i.e., device or normal vision).
- Vein Imaging Device: This within-subjects design is counter balanced for order. Each operator sees the subject's arm either initially with the normal eye or with the device, then repeats with the second condition (i.e., device or normal vision).

SUMMARY:
VueTek has developed a head mounted device that will improve the viewing of superficial, subcutaneous vasculature, differentiating it with higher contrast from surrounding tissue. Video of the vasculature is displayed to the user in a portable headset. The headset and display combination facilitates both visualization in the display and an open field of view directly to the subject's anatomy and practitioner's surroundings. The goal is to provide a non-diagnostic, enhanced visual aide that is used alongside standard visual and tactile methodology. The primary and secondary objectives of this validation are as follows:

1. Primary Objective:

   To demonstrate that the VTS1000 affords visualization of superficial, subcutaneous vascular structures, when compared to the naked eye.
2. Secondary Objective:

To demonstrate that the VTS1000 enhances visualization of superficial, subcutaneous vascular structures over the naked eye.

Validation Ancillary Endpoints

1. To gather data to demonstrate that the VTS1000 is portable, affords conventional vascular access methods, and provides flexibility, fit and balance during use.

DETAILED DESCRIPTION:
Validation methodology:

Ten (10) or more independent qualified practitioners trained to operate the device in accordance with the Directions For Use (DFU), and after completing the Device Usability aspect of the study, will be asked to perform simulated procedures with and without the device as indicated in the DFU on one-hundred (100) or more subjects using the following subject population and sampling table. A minimum of one hundred (100) or more data collection observations will be recorded, tabulated and reported.

Assumptions: The population and sampling sizes chosen for each subject category will meet the goal to attain sufficient diversity to satisfy representation that supports the efficacy of the device across the population samples. Any failures or results from the acceptance criteria may require an increase in the sampling size to ensure coverage representation of all subject demographics.

ELIGIBILITY:
1. Inclusion Criteria: All subjects will be automatically enrolled on a walk-in basis.
2. Exclusion Criteria: No walk-in subjects will be excluded from enrollment.

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Ages 4 weeks and above Light skin Dark skin Normal weight Obese weight
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To demonstrate that the VTS1000 affords visualization of superficial, subcutaneous vascular structures, when compared to the naked eye. | Immediate
  Ten (10) or more independent qualified practitioners trained to operate the device in accordance with the Directions For Use (DFU), and after completing the Device Usability aspect of the study, will be asked to perform simulated procedures with and without the device as indicated in the DFU on one-hundred (100) or more subjects using the following subject population and sampling table. A minimum of one hundred (100) or more data collection observations will be recorded, tabulated and reported.

SECONDARY OUTCOMES:
To demonstrate that the VTS1000 enhances visualization of superficial, subcutaneous vascular structures over the naked eye. | Immediate
  Ten (10) or more independent qualified practitioners trained to operate the device in accordance with the Directions For Use (DFU), and after completing the Device Usability aspect of the study, will be asked to perform simulated procedures with and without the device as indicated in the DFU on one-hundred (100) or more subjects using the following subject population and sampling table. Number of veins identified by normal vision is compared to number of veins identified with the device in a counter balanced design.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Resta-Flarer, M.D., Principal Investigator — St. Luke's Roosevelt Hospitals
Locations (1):
- St. Luke's Roosevelt Hospitals, New York, New York, United States